CLINICAL TRIAL: NCT03284645
Title: Investigating Influence of Pregnancy-induced Changes in Antiretroviral Pharmacokinetics, Together With Polymorphisms in Drug Disposition Genes, on Viral Decay Dynamics in HIV Positive Women Starting Therapy Late in Pregnancy and Postpartum
Brief Title: Viral and Antiretroviral Dynamics in HIV-1 Mother-to-Child Transmission Fluids
Acronym: VADICT
Status: Completed | Type: Observational
Sponsor: Obafemi Awolowo University (Other)
Collaborators: Federal Medical Centre, Makurdi (Unknown); University of Liverpool (Other); University of California, San Diego (Other); London School of Hygiene and Tropical Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: NHREC/01/01/2007-05/06/2017
Record Dates: First submitted 2017-09-02; First posted 2017-09-15 (Actual); Last update posted 2020-10-14 (Actual); Status verified 2020-10

CONDITIONS: Human Immunodeficiency Virus Infection
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — Tenofovir; Lamivudine; efavirenz; abacavir; Zidovudine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- ART Before or Early in Pregnancy: HIV positive pregnant women who started antiretroviral therapy (ART) before or early in pregnancy for prevention of mother-to-child transmission of HIV and for their own health.
  Interventions: Drug: Tenofovir Disoproxil Fumarate (TDF) 300 mg + Lamivudine (3TC) 300 mg + Efavirenz (EFV) 600 mg; Drug: Abacavir (ABC) 600 mg + Lamivudine (3TC) 300 mg + Efavirenz (EFV) 600 mg; Drug: Zidovudine (AZT) 300 mg + Lamivudine (3TC) 150 mg twice daily + Efavirenz (EFV) 600 mg once daily
- ART Started Third Trimester: HIV positive pregnant women starting antiretroviral therapy (ART) during the third trimester of pregnancy for prevention of mother-to-child transmission of HIV and for their own health.
  Interventions: Drug: Tenofovir Disoproxil Fumarate (TDF) 300 mg + Lamivudine (3TC) 300 mg + Efavirenz (EFV) 600 mg; Drug: Abacavir (ABC) 600 mg + Lamivudine (3TC) 300 mg + Efavirenz (EFV) 600 mg; Drug: Zidovudine (AZT) 300 mg + Lamivudine (3TC) 150 mg twice daily + Efavirenz (EFV) 600 mg once daily
- ART Started Postpartum: HIV positive women starting antiretroviral therapy (ART) after delivery for prevention of mother-to-child transmission of HIV and for their own health.
  Interventions: Drug: Tenofovir Disoproxil Fumarate (TDF) 300 mg + Lamivudine (3TC) 300 mg + Efavirenz (EFV) 600 mg; Drug: Abacavir (ABC) 600 mg + Lamivudine (3TC) 300 mg + Efavirenz (EFV) 600 mg; Drug: Zidovudine (AZT) 300 mg + Lamivudine (3TC) 150 mg twice daily + Efavirenz (EFV) 600 mg once daily

INTERVENTIONS:
Drug: Tenofovir Disoproxil Fumarate (TDF) 300 mg + Lamivudine (3TC) 300 mg + Efavirenz (EFV) 600 mg — Fixed-dose combination of 300 mg TDF, 300 mg 3TC and 600 mg EFV taken once daily.
Drug: Abacavir (ABC) 600 mg + Lamivudine (3TC) 300 mg + Efavirenz (EFV) 600 mg — Fixed-dose combination of 600 mg ABC, 300 mg 3TC and 600 mg EFV taken once daily.
Drug: Zidovudine (AZT) 300 mg + Lamivudine (3TC) 150 mg twice daily + Efavirenz (EFV) 600 mg once daily — Fixed-dose combination of 300 mg AZT and 150 mg 3TC taken twice daily, plus 600 mg EFV taken once daily.

SUMMARY:
More than 150,000 babies became infected with HIV in 2015 alone. When HIV drugs are started before or early in pregnancy, HIV positive women can give birth to HIV negative baby. This is possible because HIV drugs can reduce the amount of the virus in the body to the extent that they become undetectable by the time of delivery and during the breastfeeding period. However, some women do not start taking these drugs on time because they become infected during pregnancy or lactation. This leads to detectable virus at the time of delivery and puts the baby at risk of becoming infected. Also, the amounts of HIV drugs in the body have to be at certain levels for them to work effectively. But findings from some research have recently showed that pregnancy increases the rate at which the body removes some HIV drugs used to prevent the transfer of HIV from mother to child. While this may not cause any problem in women with no detectable virus before pregnancy, it may affect the rate at which the HIV virus is removed from the body in those starting treatment late and may put the baby at risk. This project will investigate whether the changes in drug exposure caused by pregnancy or other factors have any effect on the rate at which the HIV virus is removed from the body. HIV positive pregnant women and those who recently delivered will be recruited from different hospitals and follow up will be until breastfeeding ends. The investigators will not be involved in treatment decisions and the primary care provider will be responsible for prescribing antiretroviral regimen based on current guidelines. Samples will be collected to measure levels of the virus and the drugs in three fluids that transfer the virus to the baby: blood, genital fluid, and breastmilk. The HIV status of the babies will be monitored until they stop breastfeeding.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years old
* Planned exclusive breastfeeding until 6 months of age
* Able to understand study information and comply with follow-up schedule

Exclusion Criteria:

* Severe maternal or infant illness
* Planned exclusive formula feeding
* Taking medication with known or uncertain interaction with study drugs

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: This is cohort study of HIV positive pregnant or recently postpartum women receiving WHO recommended first-line ART regimen. Pregnant women and nursing mothers initiating ART < 4 months before delivery (n = 60) and < 6 weeks postpartum (n = 60), respectively, and a comparison group of pregnant women who initiated ART ≥ 4 months before delivery (n = 120) will be recruited from four hospitals providing PMTCT services in Nigeria.
Sampling Method: Non-Probability Sample
Enrollment: 194 (Actual)
Dates: Start 2017-12-22 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-09-17 (Actual)

PRIMARY OUTCOMES:
Polymorphisms in antiretrovirals disposition genes | At study enrolment
Minimum plasma drug concentration (Cmin) | At 2-3 months before delivery and at 10-12 weeks postpartum
Maximum plasma drug concentration (Cmax) | At 2-3 months before delivery and at 10-12 weeks postpartum
Area under the concentration-time curve (AUC) | At 2-3 months before delivery and at 10-12 weeks postpartum
Clearance over systemic availability (Cl/F) | At 2-3 months before delivery and at 10-12 weeks postpartum
HIV-1 viral load (RNA & DNA) in plasma | Through study completion (1-2 monthly)
HIV-1 viral load (RNA & DNA) in breastmilk | From 6 weeks postpartum through study completion (1-2 monthly)
HIV-1 viral load (RNA & DNA) in CVF | From week 28 to delivery (monthly)

CONTACTS AND LOCATIONS:
Overall Officials: Adeniyi Olagunju, PhD, Principal Investigator — Obafemi Awolowo University, Nigeria
Locations (4):
- Nigeria (4):
  - St. Monica's Hospital, Adikpo, Benue State
  - St. Thomas' Hospital, Ihugh, Benue State
  - Bishop Murray Medical Centre, Makurdi, Benue State
  - Federal Medical Centre, Makurdi, Benue State

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Olagunju A, Anweh D, Okafor O et al. Viral and antiretroviral dynamics in HIV mother-to-child transmission fluids (VADICT) - Protocol and data analysis plan for a cohort study [version 1; referees: awaiting peer review]. Wellcome Open Res 2019, 4:34
- [Derived] Eniayewu O, Akinloye A, Shenkoya B, Azuka U, Bolaji O, Adejuyigbe E, Owen A, Olagunju A. Prenatal efavirenz exposure is independently associated with maternal, but not fetal CYP2B6 genotype. Pharmacogenet Genomics. 2024 Oct 1;34(8):253-260. doi: 10.1097/FPC.0000000000000542. Epub 2024 Jun 24. PMID 38934229
- See also: Wellcome Open Research — https://wellcomeopenresearch.org/articles/4-34/v1